CLINICAL TRIAL: NCT04659122
Title: Phase 1b Open-label, Single Arm, Cohort Dose Escalation Study Evaluating the Safety, Tolerability, and Feasibility of Intervention With AT-100 (rhSP-D) in Intubated Patients Receiving Invasive Mechanical Ventilation With Severe COVID-19 Infection or Respiratory Failure Secondary to Severe Community Acquired Pneumonia
Brief Title: A Clinical Safety Study on AT-100 in Treating Adults With Severe COVID-19 Infection or Severed Community Acquired Pneumonia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination / study goals reached
Sponsor: Airway Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-100/002
Record Dates: First submitted 2020-12-04; First posted 2020-12-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Undefined
Keywords: COVID-19; Mechanical Ventilation; Respiratory Support; recombinant human Surfactant Protein-D (rhSP-D); Community-acquired Pneumonia; CAP; zelpultide alfa
MeSH Terms: conditions — COVID-19; Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Phase 1b portion is a dose escalation study to establish the safest & most tolerable AT-100 dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AT-100 75 mg (Experimental): Once daily AT-100 via intratracheal administration for up to 7 doses.
  Interventions: Biological: AT-100
- AT-100 150 mg (Experimental): Once daily AT-100 via intratracheal administration for up to 7 doses, if the prior dose level was safe & tolerated.
  Interventions: Biological: AT-100
- AT-100 75 mg or 150 mg (Optional Cohort) (Experimental): Once daily AT-100 via intratracheal administration for up to 7 doses, at the highest safe & tolerated dose as determined by the prior 2 dosing levels.
  Interventions: Biological: AT-100

INTERVENTIONS:
Biological: AT-100 — reconstituted AT-100 for intratracheal administration
  Other Names: (rhSP-D)

SUMMARY:
The purpose of this study is to determine if an investigational drug, AT-100, is safe and tolerated by adults who have severe corona virus disease 2019 (COVID-19) or respiratory failure secondary to severe community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is an adult ≥18 years of age.
2. The subject has documented, laboratory-confirmed SARS-CoV-2 infection within 2 weeks prior to enrollment, or meets criteria for severe community acquired pneumonia (CAP) specified in inclusion 3 below.
3. The subject has severe SARS-CoV-2 infection requiring intubation and mechanical ventilation. Or, the subject is admitted for severe CAP with respiratory failure as demonstrated by the following:

3. i. Respiratory failure requiring intubation and mechanical ventilation, and 3. ii. A clinical diagnosis of CAP that includes radiographic findings of new pulmonary infiltrate(s) consistent with CAP plus any one of the following on admission to the hospital: 3. ii. 1. Fever (Temperature > 38.0°C), 3. ii. 2. Hypothermia (Temperature < 36.0°C), 3. ii. 3. Leukocytosis with White Blood Cells (WBC) > 10,000 cells/µL or immature band forms > 10%, 3. ii. 4. Leukopenia with WBC < 4,000 cells/µL, or 3. ii. 5. Hypotension Mean Arterial Pressure (MAP) < 70 mmHg, requiring the initiation of vasopressor support.

4. The subject has been receiving mechanical ventilation for <72 hours. 5. The subject is receiving mechanical ventilation due to respiratory disease that is primarily due to SARS-CoV-2 infection or CAP.

6. The subject, or legally authorized representative if acting on the subject's behalf, is able to provide informed consent.

Exclusion Criteria:

1. The subject refuses to participate, or the subject's legally authorized representative acting on the subject's behalf refuses the subject's participation.
2. The subject is pregnant or breastfeeding.
3. The subject is anticipated to be transferred to another hospital that is not a study site within 36 hours of enrollment.
4. The subject has received or is receiving extracorporeal membrane oxygenation (ECMO) treatment for COVID-19 or CAP treatment.
5. The subject has Human Immunodeficiency virus (HIV) under highly active antiretroviral therapy (HAART).
6. The subject has cancer and is receiving chemotherapy treatment at any time during trial duration, or has received chemotherapy treatment within 30 days of trial enrollment.
7. The subject has a prior history of lung transplant, lobectomy, or other significant lung surgeries that would indicate an already compromised lung.
8. The subject has known pulmonary air leaks, such as pneumothorax and pneumomediastinum.
9. Concurrent enrollment in an investigational product, device, or treatment trial or is projected to participate in any other trial that alters the standard of care during the period of this study
10. The subject has a known allergy, sensitivity, or contraindication to any component of the test article (AT-100).
11. The subject has any active do not resuscitate (DNR)-Comfort Care (CC) order in place. Subjects with an active DNR-Comfort Care Arrest (CCA) are not excluded.
12. The subject's intubation, re-intubation, or remaining on intubation is not per clinical standard-of-care and is solely for the purposes of administration of study drug.
13. The subject has any condition or is in a situation in which, in the Investigator's judgement, puts the subject at significant risk, could confound the trial results, or may significantly interfere with the subject's trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Determining the highest-tolerated & safety-tested AT-100 dose | From time of initial AT-100 dosing until the end of the dosing period, up to 7 days
  Dose escalation of AT-100 will occur to determine the maximum dose (in mg) that produces no significant Dose Limiting Toxicities or dose-related Adverse Events (AEs).

SECONDARY OUTCOMES:
Reduction in mechanical ventilation | From mechanical ventilation initiation up to Day 28
  Days on mechanical ventilation.

OTHER OUTCOMES:
Mortality | Through study completion, up to Day 90
  Incidence of death.

CONTACTS AND LOCATIONS:
Overall Officials: Marc O. Salzberg, MD, Study Chair — Airway Therapeutics, Inc.
Locations (1):
- Airway Therapeutics Investigational Site, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Manson JJ, Crooks C, Naja M, Ledlie A, Goulden B, Liddle T, Khan E, Mehta P, Martin-Gutierrez L, Waddington KE, Robinson GA, Ribeiro Santos L, McLoughlin E, Snell A, Adeney C, Schim van der Loeff I, Baker KF, Duncan CJA, Hanrath AT, Lendrem BC, De Soyza A, Peng J, J'Bari H, Greenwood M, Hawkins E, Peckham H, Marks M, Rampling T, Luintel A, Williams B, Brown M, Singer M, West J, Jury EC, Collin M, Tattersall RS. COVID-19-associated hyperinflammation and escalation of patient care: a retrospective longitudinal cohort study. Lancet Rheumatol. 2020 Oct;2(10):e594-e602. doi: 10.1016/S2665-9913(20)30275-7. Epub 2020 Aug 21. PMID 32864628
- [Background] Sorensen GL. Surfactant Protein D in Respiratory and Non-Respiratory Diseases. Front Med (Lausanne). 2018 Feb 8;5:18. doi: 10.3389/fmed.2018.00018. eCollection 2018. PMID 29473039
- See also: Airway Therapeutics' corporate website — http://www.airwaytherapeutics.com